CLINICAL TRIAL: NCT02227420
Title: Effects of IL-1 Beta on the Hypothalamic-pituitary-adrenal (HPA) Axis in Obese Persons - the CortIL-Study
Brief Title: Effects of IL-1 Beta on the HPA-axis in Obese Persons
Acronym: CortIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EKNZ 2014-175
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome; Hypersecretion; Cortisol
MeSH Terms: conditions — Metabolic Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra (Experimental): Anakinra 100mg s.c. x 5
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra 100mg s.c. x 5

SUMMARY:
In obese individuals cortisol production and secretion is increased but the underlying mechanism is not known. Obesity leads to a pathological activation of the innate immune system partly driven by tissue production of IL-1β. Furthermore, IL-1β is also known to stimulate the release of adrenocorticotropin hormone (ACTH). Therefore, the investigators hypothesise that in obese individuals tissue inflammation stimulates ACTH via IL-1β, thereby explaining the observed hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* BMI >30kg/m2 and at least 1 manifestations of the metabolic syndrome (i.e. diabetes/ prediabetes, hypertension, dyslipidemia)
* Willingness to use contraceptive measures adequate to prevent becoming pregnant

Exclusion Criteria:

* Medication with glucocorticosteroids
* Known Cushing Syndrome
* Pregnancy or breast feeding
* Clinical signs of infection in the week before inclusion or history of a severe infection during the last 2 months
* Hematologic disease (leukocyte count < 1.5x109/l, hemoglobin <11 g/dl, platelets <100 x 103/ul)
* Kidney disease (creatinine-clearance < 30ml/min))
* Liver disease (transaminases >4x upper normal range)
* Active carcinoma
* History of tuberculosis
* Alcohol consumption >40g/d for men, >30g/d for women
* Known allergy towards anakinra
* Subject refusing or unable to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Morning cortisol levels | 14 days

SECONDARY OUTCOMES:
effect of anakinra/Kineret® on salivary cortisol, free urinary cortisol, and serum cortisol levels after an overnight dexamethasone suppression test | 14 days
correlation between the percentage of body fat or body mass index, and suppression of cortisol levels after injection of anakinra/Kineret® | 14 days
correlation between inflammatory parameters with cortisol levels | 14 days
impact of anakinra/Kineret® on other pituitary and peripheral hormones, such as: ACTH, TSH, fT4, GH, IGF-1, LH, FSH, testosterone copeptin, IL-6, CRP, leukocyte count and body temperature. | 14 days
  impact of anakinra/Kineret® on other pituitary and peripheral hormones such as: ACTH, thyroid-stimulating Hormone (TSH), free thyroxine 4 (fT4), growth Hormone (GH), insulin like growth factor (IGF)-1, luteinizing Hormone (LH), follicle stimulating Hormone (FSH), testosterone copeptin, interleukin (IL)-6, C reactive protein (CRP), leukocyte count and body temperature.
comparison of 1mg and 2mg dexamethasone suppression test | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hopsital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Urwyler SA, Ebrahimi F, Burkard T, Schuetz P, Poglitsch M, Mueller B, Donath MY, Christ-Crain M. IL (Interleukin)-1 Receptor Antagonist Increases Ang (Angiotensin [1-7]) and Decreases Blood Pressure in Obese Individuals. Hypertension. 2020 Jun;75(6):1455-1463. doi: 10.1161/HYPERTENSIONAHA.119.13982. Epub 2020 Apr 10. PMID 32275191
- [Derived] Urwyler SA, Cupa N, Christ-Crain M. Comparison of 1 mg versus 2 mg Dexamethasone Suppression Test in Patients with Obesity. Horm Metab Res. 2017 Nov;49(11):854-859. doi: 10.1055/s-0043-119128. Epub 2017 Sep 29. PMID 28962047
- [Derived] Urwyler SA, Schuetz P, Ebrahimi F, Donath MY, Christ-Crain M. Interleukin-1 Antagonism Decreases Cortisol Levels in Obese Individuals. J Clin Endocrinol Metab. 2017 May 1;102(5):1712-1718. doi: 10.1210/jc.2016-3931. PMID 28324042